CLINICAL TRIAL: NCT06980883
Title: Assessing Impact of Myofascial Release Versus Dry Needling for Chondromalacia in Adult Females: A Randomized Controlled Trial
Brief Title: Assessing Impact of Myofascial Release Versus Dry Needling for Chondromalacia in Adult Females
Acronym: females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Doaa Saeed Mohamed, lecturer at department of physical therapy for women's health, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00014233-6
Record Dates: First submitted 2025-04-28; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chondromalacia
Keywords: chondromalacia,females, myofascial release, and dry needles
MeSH Terms: conditions — Cartilage Diseases | interventions — Dry Needling; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: A total of 45 adult female diagnosed with chondromalacia and confirmed by physical examination using a patellar grind test to confirm clarke's sign were recruited for this study from the out patient clinic and soad kafafi's educational hospital , Investigations that analysed the H/Q ratio by the use of gravity corrected isokinetic strength testing
Who Masked: Investigator, Outcomes Assessor
Masking Description: double blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1:adding dry needle to traditional exercises (Experimental): Received dry needling combined with traditional treatment( straight leg raising and isometric quadriceps exercises) for 3 weeks, 2 sessions per weak.
  Interventions: Other: Dry Needling; Other: (traditional exercises)
- group 2: adding myofascial release to traditional exercises (Experimental): Myofascial Release: Provided to patients in Group 2 along with traditional treatment( 2 days per week).Evaluation of fascial restriction was assessed using the therapists elbow. Any restrictions felt were assessed and given treatment.
  Interventions: Other: myofascial release; Other: (traditional exercises)
- group 3: (control group): Applied Traditional exercise (Active Comparator): Traditional Treatment ( exercise) : Applied uniformly across all groups, comprising straight leg raising and isometric quadriceps exercises (2 days per week).
  Interventions: Other: (traditional exercises)

INTERVENTIONS:
Other: Dry Needling — dry needles Administered to patients in Group 1 as part of their treatment regimen( 2 days per week).
  Arms: group 1:adding dry needle to traditional exercises
Other: myofascial release — Myofascial Release: Provided to patients in Group 2 along with traditional treatment( 2 days per week).
  Evaluation of fascial restriction was assessed using the therapists elbow. Any restrictions felt were assessed and given treatment.Myofascial chain release- Position of the patient- Supine lying, prone lying and side lying Position of the therapist- Side of the patient limb to be treated
  - Technique-Using the therapist elbow a vertical release proximal to the attachment of the muscle belly or fascia was applied. Once an end-feel was reached a slow stroke down the length of the target tissue was performed along with monitoring the indirect feedback and tissue tension to identify any additional restrictions. The long stroke was repeated in a line parallel to the first stroke. It was continued until an end-feel is reached throughout the entire muscle belly or fascia on the most restricted/ painful points.
  Arms: group 2: adding myofascial release to traditional exercises
Other: (traditional exercises) — comprising straight leg raising and isometric quadriceps exercises (2 days per week).

SUMMARY:
Assessing Impact of Myofascial Release versus Dry Needling for Chondromalacia in Adult females. The study employed a Randomized Controlled Trial (RCT) design.

DETAILED DESCRIPTION:
A total of 45 female patients diagnosed with chondromalacia and confirmed by physical examination using a patellar grind test to confirm Clarke's sign were recruited for this study from the out patient clinic and Soad Kafafi's educational hospital , Investigations that analyzed the H/Q ratio by the use of gravity corrected isokinetic strength testing.

Inclusion criteria were:

* Age between 18-50 years old, the anterior knee pain recorded while one of the following activities at least :ascending and descending stairs, prolonged sitting and kneeling.
* Subject experiences pain during palpation of patellar facets or while performing a 25-cm step down test or double legged squat.
* Exclusion criteria included meniscal or intra-articular pathological conditions, cruciate or collateral ligaments involvement, tenderness over the patellar tendon .
* These participants were randomly assigned to one of three groups, each consisting of 15 patients all received treatment for 3 weeks, 2 sessions per weak.

Group 1: Received dry needling combined with traditional treatment( straight leg raising and isometric quadriceps exercises) for 3 weeks, 2 sessions per weak.

Group 2: Received myofascial release in addition to traditional treatment for 3 weeks, 2 sessions per week. Evaluation of fascial restriction was assessed using the therapists elbow.

Myofascial chain release:

Position of the patient: Supine lying, prone lying and side lying Position of the therapist: Side of the patient limb to be treated

-Technique: Using the therapist elbow a vertical release proximal to the attachment of the muscle belly or fascia was applied. Once an end-feel was reached a slow stroke down the length of the target tissue was performed along with monitoring the indirect feedback and tissue tension to identify any additional restrictions. The long stroke was repeated in a line parallel to the first stroke. It was continued until an end-feel is reached throughout the entire muscle belly or fascia on the most restricted/ painful points.

Traditional Treatment ( exercise) : Applied uniformly across all groups, comprising straight leg raising and isometric quadriceps exercises (2 days per week).

Group 3: Received only the traditional treatment only for 3 weeks, 2 sessions per weak.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years old, the anterior knee pain recorded while one of the following activities at least :ascending and descending stairs, prolonged sitting and kneeling.
* Subject experiences pain during palpation of patellar facets or while performing a 25-cm step down test or double legged squat. (Iiona, 2020)

Exclusion Criteria:

* excluded meniscal or intra-articular pathological conditions, cruciate or collateral ligaments involvement, tenderness over the patellar tendon .
* These participants were randomly assigned to one of three groups, each consisting of 15 patients all received treatment for 3 weaks, 2 sessions per weak.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
The isokinetic muscle strength | 3 weeks
  * Peak Torque (PT): Measured using the isokinetic dynamometer system to assess the strength of the muscles.
  * AGO/ANT Ratio: Evaluated using the isokinetic dynamometer system to examine the balance between agonist and antagonist muscle groups.
pain intensity by visual analogue scale. | 3 Weeks
  Visual Analogue Scale (VAS): Utilized to measure the intensity of pain experienced by the patients.

SECONDARY OUTCOMES:
Quality of Life physical and mental states | 3 Weeks
  Quality of Life Scale Questionnaire (QLS): Administered to assess both the physical and mental status of the patients.
Activity and functional levels of Lower Extremity | 3 weeks
  Lower Extremity Scale Questionnaire (LES): Used to evaluate the activity levels and functionality of the patients' lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa S Mohamed, lecturer, Principal Investigator — lecturer physical therapy for women health Badr University at Cairo
Locations (1):
- Masr university for sceince and technology, Cairo, Egypt